CLINICAL TRIAL: NCT00002453
Title: An Open-Label, Multicenter, Compassionate Access Study of the Safety of Tenofovir Disoproxil Fumarate Administered in Combination With Other Antiretroviral Agents for the Treatment of HIV-1 Infected Patients
Brief Title: A Compassionate Use Study of Tenofovir Disoproxil Fumarate as Treatment for HIV Infection
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Gilead Sciences (Industry)
Organization: NIH AIDS Clinical Trials Information Service (Industry)
Purpose: Treatment
Other Study IDs: 283C; GS-99-908
Record Dates: First submitted 2000-01-24; First posted 2001-08-31 (Estimated); Last update posted 2005-06-24 (Estimated); Status verified 2000-05

CONDITIONS: HIV Infections
Keywords: HIV-1; Drug Therapy, Combination; Disease Progression; Anti-HIV Agents
MeSH Terms: conditions — HIV Infections; Disease Progression | interventions — Tenofovir

INTERVENTIONS:
Drug: Tenofovir disoproxil fumarate

SUMMARY:
This study allows patients who need a new anti-HIV treatment to take tenofovir disoproxil fumarate (tenofovir DF), an experimental drug. This study also looks at any side effects the drug causes.

DETAILED DESCRIPTION:
HIV-1-infected patients who are currently receiving stable antiretroviral therapy add tenofovir DF to their regimen. Study participation lasts for approximately 48 weeks. Interested patients should contact their physicians.

ELIGIBILITY:
Inclusion Criteria

You may be eligible for this study if you:

* Are HIV-positive.
* Have a viral load greater than or equal to 10,000 copies/ml.
* Have a CD4 count less than or equal to 50 cells/mm3, or have a CD4 count greater than 50 and no more than 200 cells/mm3 with an opportunistic (AIDS-related) infection within 90 days of study entry. (Patients with a CD4 count above 200 cells/mm3 may be considered depending on drug supply.)
* Are at least 18 years old.
* Agree to use barrier methods of birth control (such as condoms) while on the study and for 30 days afterward.
* Have a life expectancy of at least one year.

Exclusion Criteria

You will not be eligible for this study if you:

* Have a history of a serious kidney or bone disease.
* Have severe nausea, vomiting, or trouble taking medications by mouth.
* Are pregnant or breast-feeding.
* Abuse alcohol or other substances that your doctor thinks would interfere with taking this medicine.
* Are taking any medicines that interfere with kidney functions.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 300
Dates: Start 1999-12

CONTACTS AND LOCATIONS:
Locations (1):
- Tenofovir Coordinating Center, Foster City, California, United States